CLINICAL TRIAL: NCT07299773
Title: Evaluation of Patients With Hypertensive Disorders of Pregnancy: An Ambispective Observational Study
Acronym: PREP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Di Pasquo Elvira, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 8162
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia; Preeclampsia (PE); Hypertensive Disorder of Pregnancy
Keywords: preeclampsia; ophtalmic nerve; ophtalmic artery
MeSH Terms: conditions — Pre-Eclampsia; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preeclamptic women > 22 weeks: All eligible patients meeting inclusion criteria during the study period will be enrolled, as no sample-size calculation is feasible due to the absence of prior literature.
  Inclusion Criteria Pregnancies complicated by preeclampsia or gestational hypertension ≥22 weeks Age ≥18 years Signed informed consent Exclusion Criteria Intrauterine fetal demise Major fetal anomalies or chromosomal abnormalities Maternal cardiac disease or ongoing cardiologic therapy Chronic kidney disease Twin or multiple pregnancies Pregestational diabetes Study Procedures
  At enrollment and near delivery, all patients will undergo:
  Non-invasive hemodynamic assessment (USCOM-1A): HR, SV, CO, TVR, inotropy index, PKR, systolic and diastolic blood pressure.
  Maternal blood testing for sFlt-1/PlGF ratio. Uterine artery Doppler: systolic peak and pulsatility index. Ophthalmic artery Doppler and ONSD measurement: performed bilaterally in supine position; PSV peaks and PSV ratio calculated.
  Carotid Doppler (CFTI): meas
  Interventions: Diagnostic Test: Doppler evaluation

INTERVENTIONS:
Diagnostic Test: Doppler evaluation — Non-invasive hemodynamic assessment (USCOM-1A): HR, SV, CO, TVR, inotropy index, PKR, systolic and diastolic blood pressure.
  Maternal blood testing for sFlt-1/PlGF ratio. Uterine artery Doppler: systolic peak and pulsatility index. Ophthalmic artery Doppler and ONSD measurement: performed bilaterally in supine position; PSV peaks and PSV ratio calculated.
  Carotid Doppler (CFTI): measured at baseline and after PLR; ΔCFTI of 10-15% considered indicative of fluid responsiveness.
  Lung ultrasound POCUS: evaluation of 8 thoracic zones using a curvilinear probe; ≥3 B-lines bilaterally considered positive for interstitial edema.

SUMMARY:
The overall objective of this study is to evaluate the prognostic role of ultrasound and laboratory parameters, specifically their potential ability to predict severe forms of preeclampsia and adverse maternal-fetal outcomes.

In particular, the aim of the present research is to obtain data on the prognostic value of ultrasonographic and biochemical parameters in patients with hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
This is an ambispective, observational cohort study conducted at a national tertiary obstetric center. This study investigates maternal hemodynamic, Doppler, ultrasound, and biochemical parameters as potential predictors of disease progression in women with gestational hypertension or preeclampsia. The study integrates non-invasive cardiovascular monitoring, placental biomarkers, ophthalmic and uterine artery Doppler velocimetry, carotid flow time index (CFTI), optic nerve sheath diameter (ONSD), and lung ultrasound.

The primary objective is to evaluate the prognostic performance of these parameters in predicting severe forms of preeclampsia and adverse maternal or perinatal outcomes. Secondary objectives include assessing the utility of lung ultrasound and carotid Doppler in characterizing maternal fluid status and supporting clinical decision-making regarding fluid management.

At enrollment and near delivery, participants undergo the following assessments:

1. Non-invasive Maternal Hemodynamics (USCOM-1A) Parameters include heart rate, stroke volume, cardiac output, total vascular resistance, inotropy index, pulse pressure, and peripheral vascular measurements. Values will be converted to Z-scores using gestational age-adjusted reference curves where applicable.
2. Placental Biomarkers Maternal blood samples are collected to determine the sFlt-1/PlGF ratio as an indicator of angiogenic imbalance.
3. Uterine Artery Doppler Uterine artery systolic peak velocities and pulsatility index are measured bilaterally using standardized transabdominal technique.
4. Ophthalmic Artery Doppler and ONSD Bilateral ophthalmic artery velocimetry is performed in a supine position to assess intracranial vascular impedance. Optic nerve sheath diameter is measured 3 mm behind the globe using a linear probe.
5. Carotid Doppler (CFTI) Carotid flow time index is measured at baseline and after a passive leg raise (PLR) maneuver. A PLR-induced ΔCFTI of 10-15% is explored as a surrogate of fluid responsiveness.
6. Lung Ultrasound (POCUS) Eight thoracic zones are evaluated using a curvilinear probe. The presence and distribution of B-lines are recorded to identify early interstitial pulmonary edema.

Clinical, obstetric, laboratory, and therapeutic data are collected longitudinally until delivery. Maternal and neonatal outcomes include timing of delivery, mode of delivery, birthweight, neonatal morbidity, and the interval between diagnosis and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies complicated by preeclampsia or gestational hypertension ≥22 weeks
* Age ≥18 years
* Signed informed consent

Exclusion Criteria:

* intrauterine fetal demise
* Major fetal anomalies or chromosomal abnormalities
* Maternal cardiac disease or ongoing cardiologic therapy
* Chronic kidney disease
* Twin or multiple pregnancies
* Pregestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: preeclamptic women > 22 weeks
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
prediction of preeclampsia with severe features | at enrollment
  Correlation between:
  hemodynamic assessment using USCOM serum levels of the biochemical markers sFlt-1/PlGF Doppler velocimetry of the uterine arteries Doppler velocimetry of the ophthalmic artery ultrasound assessment of the optic nerve sheath diameter ultrasound evaluation of carotid artery blood flow using CFTI presence of B-lines on lung ultrasound and the incidence of preeclampsia with severe features.

IPD SHARING:
Plan to Share IPD: Undecided